CLINICAL TRIAL: NCT01785329
Title: A Randomized Study of the Relative Bioavailability, Pharmacodynamics, Safety of SAR236553 (REGN727) After Single Subcutaneous Administration at 3 Different Injection Sites in Healthy Subjects
Brief Title: Pharmacokinetic of Alirocumab SAR236553 (REGN727) Administered Subcutaneously at 3 Different Injection Sites in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BDR13362; 2012-005005-40; U1111-1134-2618 (Other: UTN)
Record Dates: First submitted 2013-01-30; First posted 2013-02-07 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- alirocumab SAR236553 (REGN727) - Dose A (Experimental): alirocumab SAR236553 (REGN727) - Dose A - Injection in healthy subjects through subcutaneous administration in the abdomen.
  alirocumab SAR236553 (REGN727) is a fully human monoclonal antibody that binds PCSK9 (proprotein convertase subtilisin/kexin type 9)
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- alirocumab SAR236553 (REGN727) - Dose B (Experimental): alirocumab SAR236553 (REGN727) - Dose B - Injection in healthy subjects through subcutaneous administration in the upper arm.
  Interventions: Drug: alirocumab SAR236553 (REGN727)
- alirocumab SAR236553 (REGN727) - Dose C (Experimental): alirocumab SAR236553 (REGN727) - Dose C - Injection in healthy subjects through subcutaneous administration in the thigh.
  Interventions: Drug: alirocumab SAR236553 (REGN727)

INTERVENTIONS:
Drug: alirocumab SAR236553 (REGN727) — Pharmaceutical form:Solution for injection Route of administration: Subcutaneous

SUMMARY:
Primary Objective:

To assess the relative bioavailability of a single subcutaneous dose of alirocumab SAR236553 (REGN727) administered at 3 different injection sites in healthy subjects.

Secondary Objectives:

* To assess the pharmacodynamic effect of a single subcutaneous dose of alirocumab SAR236553 (REGN727) on serum low-density lipoprotein cholesterol and other lipids and apolipoproteins.
* To assess the safety of a single subcutaneous dose of alirocumab SAR236553 (REGN727).
* To assess the immunogenicity of a single subcutaneous dose of alirocumab SAR236553 (REGN727).

DETAILED DESCRIPTION:
Total duration of the study per subject is about 15 weeks.

ELIGIBILITY:
Inclusion criteria:

Healthy subjects.

Exclusion criteria:

Healthy subjects with history or presence of clinically relevant illness.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the serum concentrations of alirocumab SAR236553 (REGN727) after a single subcutaneous administration at 3 different injection sites in healthy subjects as a measure of the pharmacokinetics of this investigational medicinal product. | Up to 12 weeks

SECONDARY OUTCOMES:
Assessment of the serum concentrations of low-density lipoprotein cholesterol after a single subcutaneous administration of alirocumab SAR236553 (REGN727) as a measure of the pharmacodynamic effect of this investigational medicinal product. | Up to 12 weeks
Assessment of the number of subjects with adverse events after a single subcutaneous administration of alirocumab SAR236553 (REGN727) as a measure of the safety/tolerability of this investigational medicinal product. | Up to 12 weeks
Assessment of the serum concentration of anti-drug antibodies after a single subcutaneous dose of alirocumab SAR236553 (REGN727) as a measure of the immunogenicity of this investigational medicinal product. | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 826001, London, United Kingdom

REFERENCES:
- [Derived] Lunven C, Paehler T, Poitiers F, Brunet A, Rey J, Hanotin C, Sasiela WJ. A randomized study of the relative pharmacokinetics, pharmacodynamics, and safety of alirocumab, a fully human monoclonal antibody to PCSK9, after single subcutaneous administration at three different injection sites in healthy subjects. Cardiovasc Ther. 2014 Dec;32(6):297-301. doi: 10.1111/1755-5922.12093. PMID 25256660